CLINICAL TRIAL: NCT03064412
Title: Effect of Pregnancy on Androgenic Steroids in Different Genetic Panels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-145
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Sex Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Urine sample collection — A urine sample will be collected in each of the 3 trimesters of pregnancy, and also at 6 weeks post partum.
Biological: Saliva collection — A saliva sample will be collected at one time point during the study - likely at the initial baseline visit.

SUMMARY:
Androgens are important sex steroids in women. Androgens influence protein synthesis and muscle growth, are involved in maturation of the reproductive organs, have a fat reducing effect , have a negative effect on the serum lipid profile, and may also increase insulin resistance and coagulation activity. The role of androgens in women is not clear. This study is aimed at learning about the amount of androgen and its actions in pregnant women. This study is also looking to see if there are specific patient factors (such as genetics) that change the amount of androgen and its activity.

DETAILED DESCRIPTION:
There is a lot of information about the main female sex hormones such as estrogens and progesterones (the main female sex hormones and the most important in menstrual , reproductive cycles and pregnancy) . However there is little information about androgens in pregnant women. It is known that certain illnesses, chemicals and dietary products might change the amount of androgen and its actions, which could affect the mother and her baby. It is also known that there are differences between the androgen levels in different people, and in different ethnic groups. These differences are mostly due to genetic factors. The goal of this study is to learn about the androgen levels in healthy pregnant women and if genetic or clinical factors (for example age, trimester of pregnancy, parity, ethnicity, etc.) play a role in changing the androgen amount and action, throughout pregnancy and after delivery.

ELIGIBILITY:
Inclusion Criteria:

* healthy women without drug treatment, in the age range of 18-40 years

Exclusion Criteria:

* Any chronic disease such as Hypertension or Diabetes Mellitus
* Positive for HIV, hepatitis, Syphilis
* Abnormal laboratory test results (e.g. abnormal TSH, glucose, creatinine, HIV, HBV, VDRL)
* PCOS
* Ongoing hormonal treatment-e.g. progesterone, estrogen or other
* Smoking cigarettes, alcohol, regular substance use
* Confirmed or suspected abuse of drugs
* Chronic prescription drugs
* Pre-existing diabetes or GDM in last pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 70 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in sex steroids | 1st trimester (1-12 weeks gestation), 2nd trimester (13-28 weeks gestation), 3rd trimester (28-40 weeks gestation), 6 weeks post-partum
  Changes to levels of sex steroids throughout pregnancy and after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No